CLINICAL TRIAL: NCT04225039
Title: A Phase II Study of the Anti-GITR Agonist INCAGN1876 and the PD-1 Inhibitor INCMGA00012 in Combination With Stereotactic Radiosurgery in Recurrent Glioblastoma
Brief Title: Anti-GITR/Anti-PD1/Stereotactic Radiosurgery, in Recurrent Glioblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 834197
Record Dates: First submitted 2019-12-23; First posted 2020-01-13 (Actual); Results first posted 2023-09-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Immune Checkpoint Inhibitors; Radiosurgery

STUDY DESIGN:
Intervention Model Description: The overall study population will be broken down into two cohorts: Cohort A (N=16) and Cohort B (N=16). Subjects for whom surgical resection is not clinically indicated at the time of study screening will be enrolled into Cohort A (non-surgical cohort). Subjects for whom surgical resection is clinically indicated at the time of study screening will be enrolled into Cohort B (surgical cohort).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Subjects in this arm (N=16) receive a single priming dose of both INCMGA00012 (500mg) and INCAGN01876 (300mg) prior to stereotactic radiosurgery (SRS), then undergo SRS (8 Gy x 3 fractions). Following SRS, INCMGA00012 (500mg IV every 4 weeks) and INCAGN01876 (300mg IV every 2 weeks) are resumed and continued until disease progression, unacceptable toxicity, or for 2 years, whichever occurs first.
  Interventions: Drug: INCMGA00012; Drug: INCAGN01876; Drug: SRS
- Cohort B sub-arm #1 (Experimental): Subjects in this arm (N=8) receive neoadjuvant immunotherapy INCMGA00012 (500mg) + INCAGN01876 (300mg) + SRS. Subjects then undergo surgery. Postoperatively, the immunotherapy combination of INCMGA00012 (500 mg IV every 4 weeks) and INCAGN01876 (300mg IV every 2 weeks) is resumed and continued until disease progression, unacceptable toxicity, or for 2 years, whichever occurs first.
  Interventions: Drug: INCMGA00012; Drug: INCAGN01876; Drug: SRS; Procedure: Brain surgery
- Cohort B sub-arm #2 (Experimental): Subjects in this arm (N=8) receive neoadjuvant immunotherapy INCMGA00012 + INCAGN01876 (without SRS). Subjects then undergo surgery. Postoperatively, the immunotherapy combination of INCMGA00012 (IV every 4 weeks) and INCAGN01876 (IV every 2 weeks) is resumed and continued until disease progression, unacceptable toxicity, or for 2 years, whichever occurs first.
  Interventions: Drug: INCMGA00012; Drug: INCAGN01876; Procedure: Brain surgery

INTERVENTIONS:
Drug: INCMGA00012 — 500mg IV neoadjuvant treatment; 500 mg adjuvant treatment
  Other Names: PD-1 inhibitor; PD1
Drug: INCAGN01876 — 300mg IV neoadjuvant treatment; 300 mg adjuvant treatment
  Other Names: Anti-GITR agonist; GITR
Drug: SRS — administered over the course of 3 consecutive business days (8 Gy x 3 fractions, one fraction per day, total dose 24 Gy).
  Other Names: stereotactic radiosurgery
  Arms: Cohort A; Cohort B sub-arm #1
Procedure: Brain surgery — maximal safe surgical resection of the tumor.
  Arms: Cohort B sub-arm #1; Cohort B sub-arm #2

SUMMARY:
This is a phase II study of the combination of the GITR agonist monoclonal antibody INCAGN01876, the anti-PD1 monoclonal antibody INCMGA00012, and stereotactic radiosurgery (SRS) for recurrent Glioblastoma (GBM). The investigators hypothesize that the proposed regimen will be safe and stimulate a robust anti-tumor immune response and result in improved tumor responses.

DETAILED DESCRIPTION:
The study has 2 arms:

Arm A (Cohort A) is a nonsurgical arm (N=16) that will serve as the primary study cohort and evaluated for the primary study endpoint. Subjects in this arm receive a single priming dose of both INCMGA00012 and INCAGN01876 prior to stereotactic radiosurgery (SRS), then undergo SRS (8 Gy x 3 fractions). Following SRS, INCMGA00012 (IV every 4 weeks) and INCAGN01876 (IV every 2 weeks) are resumed and continued until disease progression, unacceptable toxicity, or for 2 years, whichever occurs first.

Arm B (Cohort B) is a surgical arm (N=16) that will allow for evaluation of the effects on the tumor immune microenvironment of INCMGA00012, INCAGN01876, and SRS. In order to be enrolled on this arm, subjects must have a clinical indication for surgical resection of the recurrent GBM tumor. Prior to planned surgical resection, subjects receive neoadjuvant immunotherapy (one of two possible combinations, as outlined below). Subjects then undergo surgery. Postoperatively, the immunotherapy combination of INCMGA00012 (IV every 4 weeks) and INCAGN01876 (IV every 2 weeks) is resumed and continued until disease progression, unacceptable toxicity, or for 2 years, whichever occurs first. Subjects in the surgical arm with a focus of contrast-enhancing tumor that is amenable to SRS will be assigned to surgical sub-arm #1 of Cohort B (N=8). These subjects will receive neoadjuvant INCMGA00012 + INCAGN01876 + SRS. All other subjects enrolled on Cohort B (N=8) are treated with neoadjvuant INCMGA00012 + INCAGN01876 (without SRS).

ELIGIBILITY:
Inclusion Criteria:

1. Prior histopathologically proven diagnosis of World Health Organization (WHO) grade IV glioblastoma, OR histopathologically proven diagnosis of gliosarcoma, OR molecular diagnosis of glioblastoma per c-IMPACT-NOW criteria ("diffuse astrocytic glioma, IDH-wildtype, with molecular features of glioblastoma, WHO grade IV"; this requires presence of either amplification of EGFR, whole chromosome 7 gain AND whole chromosome 10 loss, or TERT promoter mutation). Participants are eligible if the prior diagnosis was low-grade glioma and a subsequent histological diagnosis of glioblastoma was made (e.g. secondary GBM).
2. Participants must have glial tumor that is recurrent following prior first-line radiation therapy (prior dose must have been 40-75 Gy and may have been either photon or proton radiation), and must have unequivocal evidence of tumor progression by MRI scan
3. Cohort A and Sub-Arm 1 of Cohort B only: Patient must have at least one measurable (>=1cm x 1cm) contrast-enhancing tumor focus for which stereotactic radiosurgery (SRS) is clinically indicated, as determined by the Investigator, and must be able to achieve radiation target coverage without exceeding dose constraints. The contrast-enhancing target must not be larger than 4 cm in maximal diameter. Multifocal disease is allowed as long as this criterion is met

   • Sub-Arms 2 of Cohort B can have any size tumor, and the tumor does not need to be amenable to SRS
4. Cohort B (surgical) patients only: patients must be undergoing surgery that is clinically indicated as determined by their care providers
5. Tumor O-6-methylguanine-deoxyribonucleic acid (DNA) methyltransferase (MGMT) methylation status must be available from any prior GBM tumor specimen; results of routinely used methods for MGMT methylation testing (e.g. mutagenically separated polymerase chain reaction [MSPCR] or quantitative polymerase chain reaction [PCR]) are acceptable)
6. Patients may have had treatment for an unlimited number of prior relapses but must not have had prior bevacizumab or other vascular endothelial growth factor (VEGF/VEGFR) inhibitors (exception: prior bevacizumab is allowed if it was administered for the treatment of radiation necrosis rather than progressive tumor and was stopped at least 4 weeks prior to MRI showing demonstrating tumor progression). Prior gliadel wafers are only allowed if placed during the first surgery for GBM at initial diagnosis.
7. Patients must have recovered from severe toxicity of prior therapy; the following intervals from previous treatments are required to be eligible:

   * 12 weeks from completion of radiation
   * 6 weeks from a nitrosourea cytotoxic chemotherapy
   * 3 weeks from a non-nitrosourea cytotoxic chemotherapy
   * 4 weeks from any investigational (not Food and Drug Administration [FDA]-approved for glioblastoma) agents, or within a time interval less than at least 5 half-lives of the investigational agent whichever is shorter
   * 3 weeks from any major surgery, including brain surgery for recurrent tumor resection
8. If patient is on systemic corticosteroids to treat brain edema and/or brain edema-related symptoms, the dose must be 2mg of dexamethasone (or equivalent) daily or less for a minimum of 5 days prior to first dose of study drug.
9. Patients must be able to swallow oral medications
10. Age 18 or older
11. Karnofsky performance status >= 60
12. Life expectancy >3 months
13. Absolute lymphocyte count >= 500/uL
14. Adequate hepatic function within 7 days prior to start of study treatment, defined as follows

    * Total bilirubin (except patients with Gilbert's Syndrome, who are eligible for the study but exempt from the total bilirubin eligibility criterion) ≤ 2.0 mg/dl
    * ALT and AST ≤ 2.5x upper limit of normal (ULN)
15. Adequate renal function within 7 days prior to start of study treatment, defined as follows:

    • Serum creatinine <=1.5 x institutional ULN OR calculated creatinine clearance (glomerular filtration rate can also be used in place of creatinine or CrCl) >=50 mL/min for subjects with creatinine levels >1.5x institutional ULN
16. Reproductive Status

    1. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to the start of study drug.
    2. Women must agree to not breastfeed during the study or for 180 days after the last dose of study treatment
    3. WOCBP must agree to use an adequate method to avoid pregnancy (as defined below) from the time of study screening through 180 days from last dose of study drug
    4. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception (as defined below) starting with the first dose of study drug through 180 days after the last dose of study
    5. Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, these WOCBP must still undergo pregnancy testing as described in this section.

    At a minimum, participants of childbearing potential who are sexually active and their partners must agree to the use of a highly effective form of contraception (as defined below) throughout their participation beginning with the time of consent, during the study treatment, and for 180 days after last dose of study treatment(s).

    HIGHLY EFFECTIVE METHODS OF CONTRACEPTION:
    * Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants and intrauterine devices (IUDs) by WOCBP subject or male subject's WOCBP partner. Female partners of male subjects participating in the study may use hormone-based contraceptives as one of the acceptable methods of contraception since they will not be receiving study drug
    * Nonhormonal IUDs
    * Bilateral Tubal ligation
    * Vasectomy
    * Sexual Abstinence

      * It is not necessary to use any other method of contraception when complete abstinence is elected.
      * WOCBP participants who choose complete abstinence must continue to have pregnancy tests.
      * Acceptable alternate methods of highly effective contraception must be discussed in the event that the WOCBP participants chooses to forego complete abstinence.
17. Participant must, in the opinion of the Investigator, be able to comply with study procedures
18. Patients must be able to understand the study procedures and agree to participate in the study by providing written informed consent (or have legally authorized representative sign on patient's behalf if patient physically unable to sign consent due to neurologic deficit)

Exclusion Criteria

Any of the following would exclude the subject from participation in the study:

1. Contrast-enhancing tumor in brainstem or spinal cord (subjects do not need spinal MRI for screening, but known spinal cord tumor is exclusionary)
2. Diffuse leptomeningeal disease
3. Prior bevacizumab or other vascular endothelial growth factor (VEGF/VEGFR) inhibitors (exception: prior bevacizumab is allowed if it was administered for the treatment of radiation necrosis rather than progressive tumor and was stopped at least 4 weeks prior to MRI showing demonstrating tumor progression).
4. Patients with clinically significant mass effect or midline shift (e.g., 1-2 cm of midline shift)
5. Use of any immunosuppressive medication other than steroids, including but not limited to antimetabolites, calcineurin inhibitors, and/or anti-TNF agents within six months of start of study drug
6. Prior diagnosis of immunodeficiency
7. Prior solid organ or bone marrow transplantation
8. Autoimmune or connective tissue disease that is EITHER (a) actively flaring OR (b) has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).

   EXCEPTIONS: Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, adrenal insufficiency requiring only replacement dose corticosteroids, skin disorders (such as vitiligo, psoriasis, pemphigus, or alopecia) controlled with topical medications, or conditions not expected to recur in the absence of an external trigger are permitted to enroll. Patients with asthma that is not actively flaring are allowed. Patients with history of Grave's disease that is previously treated with thyroidectomy or radioiodine are allowed. Patients with celiac disease whose symptoms are controlled with a gluten-free diet are allowed. Patients with rheumatoid arthritis and other arthropathies such as ankylosing spondylitis, Sjogren's syndrome, Raynaud syndrome, and patients with positive serologies, such as antinuclear antibodies (ANA) or anti-thyroid antibodies, should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible.
9. History of non-infectious pneumonitis that required steroid treatment
10. Known active hepatitis B virus (HBsAg reactive) or active hepatitis C virus (HCV RNA detectable by PCR)
11. Human immunodeficiency virus (HIV)-positive patients on antiretroviral therapy
12. Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen are excluded from this trial. Otherwise, patients with prior or concurrent malignancy are eligible.
13. Any serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection that, in the opinion of the investigator, would put the subject at undue risk from the study treatment.
14. Patients with uncontrolled or significant cardiovascular disease including, but not limited to, any of the following are ineligible:

    * Myocardial infarction or uncontrolled angina within 90 days prior to consent
    * History of clinically significant arrhythmia (such as ventricular tachycardia, ventricular fibrillation, or torsades pointes)
    * History of cardiomyopathy, pericarditis, significant pericardial effusion, myocarditis, or New York Heart Association (NYHA) functional class III-IV congestive heart failure
15. Known hypersensitivity to another monoclonal antibody that cannot be controlled with standard measures (e.g., antihistamines and corticosteroids)
16. Prisoners or subjects who are involuntarily incarcerated
17. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness
18. Pregnant women are excluded
19. Received a live vaccine within 30 days prior to first dose of study drug. Examples include but are not limited to measles, mumps, rubella, varicella/zoster, yellow fever, rabies, Bacillus Celmette-Guerin (BCG), and typhoid. Intranasal influenza vaccines are not allowed.
20. Participant must not be simultaneously enrolled in any interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2029-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bagley, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 39 participants signed consent. A total of 5 participants either failed to meet eligibility requirements or withdrew consent.
  A total of 18 participants were assigned to Cohort A. Because of a protocol deviation, the data of 2 participants was not used for efficacy analysis, but it was used for safety.
  A total of 8 participants were assigned to Cohort B Sub-arm #1. A total of 8 participants were assigned to Cohort B Sub-arm #2.
Groups:
- Cohort A: Subjects in this arm (N=18) receive a single priming dose of both INCMGA00012 (500mg) and INCAGN01876 (300mg) prior to stereotactic radiosurgery (SRS), then undergo SRS (8 Gy x 3 fractions). Following SRS, INCMGA00012 (500mg IV every 4 weeks) and INCAGN01876 (300mg IV every 2 weeks) are resumed and continued until disease progression, unacceptable toxicity, or for 2 years, whichever occurs first. Because of a protocol deviation, two subjects' data is not analyzed for efficacy.
  INCMGA00012: 500mg IV neoadjuvant treatment; 500 mg adjuvant treatment
  INCAGN01876: 300mg IV neoadjuvant treatment; 300 mg adjuvant treatment
  SRS: administered over the course of 3 consecutive business days (8 Gy x 3 fractions, one fraction per day, total dose 24 Gy).
- Ineligible or Withdrew Consent: Subjects in this arm (N=5) signed the consent form but were either ineligible for the study or withdrew consent and were never treated
Period: Overall Study
Arm/Group | Cohort A | Cohort B Sub-arm #1 | Cohort B Sub-arm #2 | Ineligible or Withdrew Consent
Started | 18 | 8 | 8 | 5
Completed | 15 | 7 | 8 | 0
Not Completed | 3 | 1 | 0 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Not completed — Currently active on study treatment | 0 | 1 | 0 | 0
Not completed — Protocol deviation; data not analyzed for efficacy | 2 | 0 | 0 | 0
Not completed — Ineligible for treatment | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- GITR + PD1, SRS (Cohort A): Subjects in this arm (N=18) receive a single priming dose of both INCMGA00012 (500mg) and INCAGN01876 (300mg) prior to stereotactic radiosurgery (SRS), then undergo SRS (8 Gy x 3 fractions). Following SRS, INCMGA00012 (500mg IV every 4 weeks) and INCAGN01876 (300mg IV every 2 weeks) are resumed and continued until disease progression, unacceptable toxicity, or for 2 years, whichever occurs first. Because of a protocol deviation, two subjects' data is not analyzed for efficacy.
  INCMGA00012: 500mg IV neoadjuvant treatment; 500 mg adjuvant treatment
  INCAGN01876: 300mg IV neoadjuvant treatment; 300 mg adjuvant treatment
  SRS: administered over the course of 3 consecutive business days (8 Gy x 3 fractions, one fraction per day, total dose 24 Gy).
- GITR + PD1, SRS, Surgery (Cohort B Sub-arm #1): Subjects in this arm (N=8) receive neoadjuvant immunotherapy INCMGA00012 (500mg) + INCAGN01876 (300mg) + SRS. Subjects then undergo surgery. Postoperatively, the immunotherapy combination of INCMGA00012 (500 mg IV every 4 weeks) and INCAGN01876 (300mg IV every 2 weeks) is resumed and continued until disease progression, unacceptable toxicity, or for 2 years, whichever occurs first.
  INCMGA00012: 500mg IV neoadjuvant treatment; 500 mg adjuvant treatment
  INCAGN01876: 300mg IV neoadjuvant treatment; 300 mg adjuvant treatment
  SRS: administered over the course of 3 consecutive business days (8 Gy x 3 fractions, one fraction per day, total dose 24 Gy).
  Brain surgery: maximal safe surgical resection of the tumor.
- GITR + PD1, Surgery (Cohort B Sub-arm #2): Subjects in this arm (N=8) receive neoadjuvant immunotherapy INCMGA00012 + INCAGN01876 (without SRS). Subjects then undergo surgery. Postoperatively, the immunotherapy combination of INCMGA00012 (IV every 4 weeks) and INCAGN01876 (IV every 2 weeks) is resumed and continued until disease progression, unacceptable toxicity, or for 2 years, whichever occurs first.
  INCMGA00012: 500mg IV neoadjuvant treatment; 500 mg adjuvant treatment
  INCAGN01876: 300mg IV neoadjuvant treatment; 300 mg adjuvant treatment
  Brain surgery: maximal safe surgical resection of the tumor.
- Total: Total of all reporting groups
Arm/Group | GITR + PD1, SRS (Cohort A) | GITR + PD1, SRS, Surgery (Cohort B Sub-arm #1) | GITR + PD1, Surgery (Cohort B Sub-arm #2) | Ineligible or Withdrew Consent | Total
Number analyzed (Participants) | 18 | 8 | 8 | 5 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 1 | 4 | 2 | 18
  >=65 years | 7 | 7 | 4 | 3 | 21
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [52 to 66] | 64 [63 to 65] | 63 [55 to 72] | 67 [53 to 79] | 64 [55 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 3 | 4 | 19
  Male | 10 | 4 | 5 | 1 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 2
  White | 18 | 8 | 6 | 5 | 37
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 8 | 8 | 5 | 39

OUTCOME MEASURES:

1. Primary Outcome: Objective Radiographic Response (ORR)
Description: Per modified response assessment in neuro-oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=50% decrease in the sum of the products of the perpendicular diameters of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 26 months
Population: Per protocol, it was pre-specified to only include subjects in Cohort A and the subject must have received at least one dose of BOTH study drugs AND has received at least one fraction of SRS. Because of a protocol deviation, the data of 2 subjects is not included for efficacy analysis.
Measure: Number (95% Confidence Interval); unit: % of participants with response
Arm/Group | GITR + PD1, SRS (Cohort A)
Number analyzed (Participants) | 16
% of participants with response | 0 [0 to 19]

2. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events as Assessed by NCI CTCAE v 5.0
Description: Adverse events will be evaluated by monitoring frequency, duration, and severity of adverse events (AEs) per NCI CTCAE v 5.0
Time Frame: 25 months
Reporting Status: Not Posted

3. Secondary Outcome: Overall Survival
Description: OS, defined as the time from date of enrollment until death from any cause
Time Frame: 84 months
Reporting Status: Not Posted

4. Secondary Outcome: Progression Free Survival
Description: PFS, defined as the time from date of enrollment until the earliest date of disease progression (as determined by modified RANO criteria) or death due to any cause
Time Frame: 84 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 26 months
Description: All subjects who sign informed consent will be included in safety analyses and in calculation of the rate of AEs, regardless of whether and how much study drug was received. Subjects who were determined to be ineligible for treatment or who withdrew consent and did not receive treatment are included in the safety analyses, in the "Ineligible or Withdrew Consent" cohort.
Groups:
- Cohort A: Subjects in this arm (N=18) signed the consent form and received a single priming dose of both INCMGA00012 (500mg) and INCAGN01876 (300mg) prior to stereotactic radiosurgery (SRS), then undergo SRS (8 Gy x 3 fractions). Following SRS, INCMGA00012 (500mg IV every 4 weeks) and INCAGN01876 (300mg IV every 2 weeks) are resumed and continued until disease progression, unacceptable toxicity, or for 2 years, whichever occurs first.
  INCMGA00012: 500mg IV neoadjuvant treatment; 500 mg adjuvant treatment
  INCAGN01876: 300mg IV neoadjuvant treatment; 300 mg adjuvant treatment
  SRS: administered over the course of 3 consecutive business days (8 Gy x 3 fractions, one fraction per day, total dose 24 Gy).
- Cohort B Sub-arm #1: Subjects in this arm (N=8) signed the consent form and received neoadjuvant immunotherapy INCMGA00012 (500mg) + INCAGN01876 (300mg) + SRS. Subjects then undergo surgery. Postoperatively, the immunotherapy combination of INCMGA00012 (500 mg IV every 4 weeks) and INCAGN01876 (300mg IV every 2 weeks) is resumed and continued until disease progression, unacceptable toxicity, or for 2 years, whichever occurs first.
  INCMGA00012: 500mg IV neoadjuvant treatment; 500 mg adjuvant treatment
  INCAGN01876: 300mg IV neoadjuvant treatment; 300 mg adjuvant treatment
  SRS: administered over the course of 3 consecutive business days (8 Gy x 3 fractions, one fraction per day, total dose 24 Gy).
  Brain surgery: maximal safe surgical resection of the tumor.
- Cohort B Sub-arm #2: Subjects in this arm (N=8) signed the consent form and received neoadjuvant immunotherapy INCMGA00012 + INCAGN01876 (without SRS). Subjects then undergo surgery. Postoperatively, the immunotherapy combination of INCMGA00012 (IV every 4 weeks) and INCAGN01876 (IV every 2 weeks) is resumed and continued until disease progression, unacceptable toxicity, or for 2 years, whichever occurs first.
  INCMGA00012: 500mg IV neoadjuvant treatment; 500 mg adjuvant treatment
  INCAGN01876: 300mg IV neoadjuvant treatment; 300 mg adjuvant treatment
  Brain surgery: maximal safe surgical resection of the tumor.
Arm/Group | Cohort A | Cohort B Sub-arm #1 | Cohort B Sub-arm #2 | Ineligible or Withdrew Consent
All-Cause Mortality (participants affected / at risk) | 12/18 | 0/8 | 6/8 | 4/5
Serious Adverse Events (participants affected / at risk) | 8/18 | 5/8 | 5/8 | 1/5
Other Adverse Events (participants affected / at risk) | 18/18 | 8/8 | 8/8 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=18) | Cohort B Sub-arm #1 (N=8) | Cohort B Sub-arm #2 (N=8) | Ineligible or Withdrew Consent (N=5)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalitis infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Shunt malfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema cerebral (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness left-sided (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness right-sided (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=18) | Cohort B Sub-arm #1 (N=8) | Cohort B Sub-arm #2 (N=8) | Ineligible or Withdrew Consent (N=5)
Anemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 1 (2) | 0 (0)
Other: Enlarged lymph node (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Other: Ectopic beat (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Other: Ear fullness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Other: Whooshing sound in ears (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other: Allergies (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other: Change in vision, non-specific, not blurring not diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other: Decreased ROM (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other: Double vision (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Periorbital edema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision decreased (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distention (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 2 (3) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (3) | 1 (1) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (4) | 2 (2) | 0 (0)
Other: Bright red blood in stool (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Other: Tooth sensitivity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 6 (6) | 2 (3) | 3 (3) | 0 (0)
Fatigue (General disorders) | 11 (25) | 7 (8) | 6 (9) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Generalized edema (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other: Generalized weakness (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Other: Motion sickness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Other: Coronavirus (Not SARS-CoV-2) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other: COVID 19 positive (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Other: Rash (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Other: Yeast vaginitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shingles (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (3) | 3 (3) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 6 (10) | 5 (5) | 2 (3) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Other: Broken L toe (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other: Left foot injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other: Pain, left hip, intermittent (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other: Pain, surgical incision (Injury, poisoning and procedural complications) | 1 (1) | 5 (7) | 1 (1) | 0 (0)
Other: Soft tissue inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (4) | 2 (4) | 4 (10) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (9) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 4 (7) | 1 (2) | 1 (1) | 0 (0)
Weight Loss (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 2 (8) | 1 (1) | 1 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 3 (4) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 4 (4) | 2 (2) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other: Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other: Vitamin B12 deficiency (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 2 (3) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Other: Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (3) | 1 (1) | 0 (0)
Other: Pilonidal cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 3 (5) | 1 (1) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 5 (6) | 5 (11) | 1 (2) | 0 (0)
Concentration impairment (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 3 (4) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 2 (2) | 3 (9) | 4 (6) | 0 (0)
Edema cerebral (Nervous system disorders) | 6 (7) | 2 (2) | 2 (2) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 11 (18) | 4 (7) | 3 (7) | 0 (0)
Hypoglossal nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Memory impairment (Nervous system disorders) | 8 (8) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness left-sided (Nervous system disorders) | 5 (6) | 4 (8) | 3 (5) | 0 (0)
Muscle weakness right-sided (Nervous system disorders) | 1 (2) | 3 (5) | 1 (2) | 0 (0)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other: Balance impairment (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Other: Bell's palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other: Decreased dexterity left hand (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other: Head heaviness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other: Malignant neoplasm progression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other: Neglect left-sided (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Other: Neglect right-sided (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other: Nerve pain of the face (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other: Pseudomeningocele (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Other: Tumor inflammation (Nervous system disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Other: Visual field deficit (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 3 (6) | 1 (2) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 4 (8) | 1 (1) | 3 (4) | 0 (0)
Spasticity (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 2 (3) | 4 (4) | 0 (0)
Delerium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (5) | 1 (1) | 2 (3) | 0 (0)
Other: Changes in mood, emotional (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other: Lack of motivation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Other: Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 3 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Other: Chest tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Body odor (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other: Bug bites on extremities (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other: Circular red spots (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other: Erythematous ecchymotic rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other: Milaria rubra rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other: Nodule L hand (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other: Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other: Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Other: Pustule (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Other: Rash, erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other: Skin tear (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other: Surgical incision (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 4 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (6) | 2 (2) | 1 (2) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT04225039/Prot_SAP_002.pdf
  • Informed Consent Form (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT04225039/ICF_001.pdf